CLINICAL TRIAL: NCT02433821
Title: Effectiveness of Pilates to Treat Mechanical Neck Pain
Brief Title: Pilates to Treat Neck Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luciana de Araujo Cazotti, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP_UNIFESP-0208/11
Record Dates: First submitted 2013-04-08; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Mechanical Neck Pain
Keywords: Mechanical Neck Pain; Pain; Function; Quality of life; Pilates
MeSH Terms: conditions — Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilates Group (Experimental): The group will realize 2 classes per week, lasting one our, of Pilates under supervision of a trained instructor. The training program will last 3 months.
  Interventions: Other: Pilates
- Control group (No Intervention): The patients will keep the drug treatment and will be keep in a waiting list. After the 180 days of study the will be invited to realize the Pilates training.

INTERVENTIONS:
Other: Pilates
  Arms: Pilates Group

SUMMARY:
The neck pain comes from disturbances related to the cervical spine, of multifactorial origin and is considered a frequent problem of disability.

Pilates is a physical conditioning method that has been widely used to improve posture and develop body awareness.

The aim of this study is to assess the impact of the Pilates method in the control of pain, function and quality of life in patients with chronic mechanical neck pain.

Methods: 64 patients with chronic mechanical neck pain will be selected and randomized into two groups: intervention and control. Both groups will be assessed for pain, function, quality of life and medication intake.

The intervention group will hold Pilates sessions for three months, with two sessions per week. The control group will continue with the usual drug treatment. Both groups will be instructed to use 750mg acetaminophen every 6 hours if there is pain, but consumption of the drug will be controlled.

Although the symptoms of neck pain are common in the population, no study has investigated the effects of the Pilates method as a possible treatment for neck pain. The hypothesis is that the Pilates method can offer benefits to these patients.

ELIGIBILITY:
Inclusion Criteria:

* People with diagnosis of chronic mechanical neck pain and symptoms of pain in the lower region of spine, between the occipital and the first thoracic vertebra, for more than three months.
* Pain between 3 and 8 on the numerical pain scale
* Age between 18 and 65
* Both genders
* Agree to take part in the study and sign the terms of agreement

Exclusion Criteria:

* Fibromyalgia
* Previous traumatic injuries in the spine
* Infections and inflammation in the spine cervical pain radiating to upper limbs
* The practice of physical activity started or altered in the last 3 months
* Visual deficiency not corrected by glasses, disturbance in the central nervous system, hearing deficiency making the use of the method impossible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in pain | Baseline, after 45, 90 and 180 days
  Evaluated by visual analogue scale (VAS) from 0 to 10

SECONDARY OUTCOMES:
Change in function | Baseline, after 45, 90 and 180 days
  Evaluated by the Neck Disability Index (score ranges from 0 to 50)
Change in Quality of life | Baseline, after 45, 90 and 180 days
  Evaluated by the short form 36 (SF-36) questionnaire
Change in medication intake | After 45, 90 and 180 days from baseline
  Patients fill out a specific form regarding the medication intake

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Araujo Cazotti L, Jones A, Roger-Silva D, Ribeiro LHC, Natour J. Effectiveness of the Pilates Method in the Treatment of Chronic Mechanical Neck Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Sep;99(9):1740-1746. doi: 10.1016/j.apmr.2018.04.018. Epub 2018 May 9. PMID 29752907